CLINICAL TRIAL: NCT02247440
Title: Response to Peg-interferon and Ribavirin for the Treatment of HCV Infection in HIV Co-infected Patients, Implemented in Public Hospitals in Thailand
Brief Title: HCV-HIV Co-infected Patient Cohort in Thailand
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Ministry of Health, Thailand (Other Government)
Responsible Party: Principal Investigator, GONZAGUE JOURDAIN, Researcher, Institut de Recherche pour le Developpement
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHPT-HCV
Record Dates: First submitted 2014-09-09; First posted 2014-09-25 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-02

CONDITIONS: Hepatitis C Infection; HIV
Keywords: HCV; HIV; Thailand; pegylated interferon; ribavirin
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PegINF-ribavirin (Experimental): Peg-interferon + ribavirin under HIV physician supervision Peg-interferon alpha 2-b initial dosing is 1.5 micrograms/kg (subcutaneous injection) once a week
  Ribavirin initial dosing in the morning and in the evening:
  1. For genotypes 2, 3: ribavirin 400 mg (i.e. 800 mg daily).
  2. For genotypes 1, 4, 5 and 6:
     * 800 mg/day, if bodyweight <65 kg,
     * 1000 mg/day, if bodyweight between 66-80 kg,
     * 1200 mg/day, if bodyweight between 81-105 kg,
     * 1400 mg/day, if bodyweight >105 kg.
  Duration: 48 weeks
  Interventions: Drug: Peg-interferon + ribavirin under HIV physician supervision

INTERVENTIONS:
Drug: Peg-interferon + ribavirin under HIV physician supervision — Peg-interferon + ribavirin under HIV physician supervision
  Other Names: Pegintron, Rebetol

SUMMARY:
This is a study of HCV treatment using the standard regimen of pegylated-interferon plus ribavirin in HIV co-infected patients participating in the PHPT cohort study. The treatment will be implemented in conjunction with gastro-enterologists/hepatologists by internists responsible for the participant's HIV treatment.

Chronic hepatitis C virus (HCV) infection is responsible for several severe and life threatening complications, which are worsened by HIV co-infection. HIV-HCV co-infected patients are at a higher risk of death compared to HIV mono-infected individuals, even if HIV replication is suppressed on antiretroviral treatment.

The goal of HCV antiviral treatment is to cure HCV infection. Curing HCV infection allows fibrosis regression, improved clinical outcomes. In addition, individuals who have been cured are no longer contagious to other individuals, therefore widespread access to HCV treatment may contribute to the control of the HCV epidemic.

A combination of injectable pegylated-interferon with oral ribavirin is currently the recommended regimen for the treatment of hepatitis C in the setting of HIV co-infection. They are administered for 24 weeks in HCV mono-infected patients but need to be administered for one year in HIV-HCV co-infected patients. Newer drugs, such as the first generation HCV protease inhibitors (boceprevir, telaprevir), administered concomitantly, are used in patients who have not been cured using peg-interferon + ribavirin, and may allow for shorter treatment.

PRIMARY OBJECTIVE

1. To determine the percentage of patients according to genotypes with sustained virological response 6 months after treatment discontinuation (SVR).

HCV TREATMENT

* Peg-interferon alpha 2-b (a subcutaneous injection of 1.5 micrograms/kg once a week)
* Ribavirin dosing according to HCV genotype and body weight; dose adjustment in case of anemia.

A total of 60 patients could be enrolled in the study: 15 HCV-HIV co-infected patients in a first part (starting in August 2014) and 45 patients in a second part, depending on funding.

DETAILED DESCRIPTION:
Study Population Screening: HIV infected patients with a positive anti-HCV test will be approached for screening if they are at least 18 years old, participate in the PHPT cohort study, have evidence of control of HIV replication and have a CD4 cell count ≥200 cells/mm3 if currently receiving antiretroviral HIV treatment (on the same anti-HIV regimen for at least 12 weeks); or HIV RNA load ≤5000 copies/ml CD4 cells ≥500 cells/mm3if not receiving antiretroviral treatment.

Inclusion Criteria

* Evidence of chronic HCV infection for at least 6 months before study entry (at least one detectable HCV viral load, i.e. ≥17 IU/mL, with an antibody test positive at least 6 months before the HCV RNA load result)
* Fibrosis Stage F2-3-4 determined by transient elastography (Fibroscan or other similar equipment). During the first part of the study, priority will be given to patients with Fibrosis Stage F2-3.
* Negative pregnancy test (on the day of inclusion). Main exclusion criteria
* Anemia and thrombocytopenia
* Severe liver damage, advanced stage cirrhosis or cancer
* Uncontrolled diabetes, Uncontrolled thyroid dysfunction
* Retinopathy
* Creatinine clearance <50 mL/min (Cockcroft)
* Disease associated with the immune system
* Significant heart problems
* Severe neuropsychiatric conditions
* Contra-indication to study treatment (including pregnancy or lack of effective contraception in the participant or female partner)
* Other exclusion criteria related to the use of ribavirin and peg-interferon
* Any conditions that, in the investigator's judgment, may compromise the follow up.

Follow up After HCV treatment initiation, patients will be monitored for safety and antiviral efficacy at 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44 and 48 weeks (end of treatment) and 6 months after treatment discontinuation.

Treatment will be discontinued earlier in patients who do not achieve early viral response, i.e. a decrease of at least 2 log10 HCV RNA IU/mL after the first 12 weeks of HCV therapy.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of chronic HCV infection for at least 6 months before study entry (at least one detectable HCV viral load, i.e. ≥17 IU/mL, with an antibody test positive at least 6 months before the HCV RNA load result)
* Fibrosis Stage F2-3-4 determined by transient elastography (Fibroscan or other similar equipment). During the first part of the study, priority will be given to patients with Fibrosis Stage F2-3.
* Negative pregnancy test (on the day of inclusion).

Exclusion Criteria:

* Anemia and thrombocytopenia
* Severe liver damage, advanced stage cirrhosis or cancer
* Uncontrolled diabetes, Uncontrolled thyroid dysfunction
* Retinopathy
* Creatinine clearance <50 mL/min (Cockcroft)
* Disease associated with the immune system
* Significant heart problems
* Severe neuropsychiatric conditions Contra-indication to study treatment (including pregnancy or lack of effective contraception in the participant or female partner)
* Other exclusion criteria related to the use of ribavirin and peg-interferon
* Any conditions that, in the investigator's judgment, may compromise the follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-08; Primary Completion 2017-05 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gonzague Jourdain, MD, PhD, Principal Investigator — Institut de Recherche pour le Developpement
Locations (5):
- Thailand (5):
  - Sanpatong Hospital, San Pa Tong, Chiang Mai
  - Nakornping Hospital, Chiang Mai
  - Chiangrai Prachanukroh Hospital, Chiang Rai
  - Chonburi Hospital, Chon Buri
  - Samutsakhon Hospital, Samut Sakhon

RESULTS

PARTICIPANT FLOW:
Groups:
- PegINF-ribavirin: Peg-interferon + ribavirin under HIV physician supervision Peg-interferon alpha 2-b initial dosing is 1.5 micrograms/kg (subcutaneous injection) once a week
  Ribavirin initial dosing in the morning and in the evening:
  1. For genotypes 2, 3: ribavirin 400 mg (i.e. 800 mg daily).
  2. For genotypes 1, 4, 5 and 6:
     * 800 mg/day, if bodyweight <65 kg,
     * 1000 mg/day, if bodyweight between 66-80 kg,
     * 1200 mg/day, if bodyweight between 81-105 kg,
     * 1400 mg/day, if bodyweight >105 kg.
  Duration: 48 weeks
  Peg-interferon + ribavirin under HIV physician supervision: Peg-interferon + ribavirin under HIV physician supervision
Period: Overall Study
Arm/Group | PegINF-ribavirin
Started | 18
Completed | 14
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Arm/Group | PegINF-ribavirin
Number analyzed (Participants) | 18
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 44.2 [39.6 to 51.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 18
Region of Enrollment [Number; unit: participants]
  Thailand | 18
Body Mass Index [Median (Inter-Quartile Range); unit: kg/m^2] | 21.8 [20.6 to 25.7]
HCV RNA [Median (Inter-Quartile Range); unit: log10 IU/mL] | 5.83 [5.59 to 6.75]
HCV genotypes [Count of Participants; unit: Participants] — Response to and duration of peg-interferon treatment vary according to Hepatitis C virus (HCV) genotypes. Prior to initiating HCV treatment, HCV genotype was determined using the INNO-LiPA technique.
  Participants
    Gt 1a | 2
    Gt 1b | 8
    Gt 3a | 5
    Gt 3b | 1
    Gt 6a/b | 1
    Gt 6c-l | 1
IL 28B polymorphism [Count of Participants; unit: Participants] — Single nucleotide polymorphisms (SNP) on IL-28B in particular at position called rs12979860, are associated with different responses to peg-interferon+ribavirin treatment. For example the rs12979860 CC is predictive of good response to treatment. This SNP was assessed in all participants at baseline using SNP real-time PCR assay.
  Participants
    CC | 14
    CT | 4
Liver fibrosis stage [Count of Participants; unit: Participants] — Assessment of Liver fibrosis stages is needed to decide the HCV treatment.
  Liver Fibrosis stage was assessed by transient elastography ultrasound based technique that measured the stiffness of the liver. There are five stages starting from F0 no scarring until F4: cirrhosis or advanced scarring and treatment in this study was initiated in participants with F2-F4 fibrosis stages. Response to treatment was expected to be better in participants with lower fibrosis stages.
  Participants
    F2 | 1
    F3 | 4
    F4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Virological Response 6 Months After Treatment Discontinuation
Description: Number of Participants with Sustained Virological Response 6 Months After Treatment Discontinuation,
Time Frame: 6 months after end of treatment, i.e. 1.5 years after treatment initiation
Measure: Count of Participants; unit: Participants
Arm/Group | PegINF-ribavirin
Number analyzed (Participants) | 18
Participants | 10

2. Secondary Outcome: Number of Participants With at Least a Serious Adverse Events Associated With Study Treatment (Peg-interferon and Ribavirin)
Description: Number of participants with at least a serious adverse events associated with study treatment (peg-interferon and ribavirin).
Time Frame: From initiation of treatment to 6 months after treatment discontinuation
Measure: Count of Participants; unit: Participants
Arm/Group | PegINF-ribavirin
Number analyzed (Participants) | 18
Participants | 1

3. Secondary Outcome: Number of Participants Grouped by HIV-1 RNA Concentrations
Description: Number of participants grouped by HIV-1 RNA concentrations (Detected vs. Not Detected).
Time Frame: At time of treatment discontinuation (whatever its date) and 6 months thereafter
Measure: Count of Participants; unit: Participants
Arm/Group | PegINF-ribavirin
Number analyzed (Participants) | 18
Participants
  HIV-1 RNA not detected | 16
  HIV-1 RNA detected | 1
  Missing | 1

4. Other Pre Specified Outcome: Number of Participants Completed the First 24 and 48 Weeks of Treatment
Description: Number of participants completed the first 24 and 48 weeks of treatment.
Time Frame: From initiation of treatment to the first 48 weeks of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | PegINF-ribavirin
Number analyzed (Participants) | 18
Participants
  Completed the first 24 weeks of treatment | 14
  Completed the first 48 weeks of treatment | 14

5. Other Pre Specified Outcome: Number of Adverse Events by Severity Grade
Description: Number of adverse events (AE) by severity grade. The severity grading scale is based on the DAIDS grading table, the grading scale ranging from grades 1 to 5: Grade 1 indicates a mild event, Grade 2 indicates a moderate event, Grade 3 indicates a severe event, Grade 4 indicates a potentially life-threatening event, and Grade 5 indicates death.
Time Frame: From initiation of treatment to 6 months after treatment discontinuation
Measure: Number; unit: events
Arm/Group | PegINF-ribavirin
Number analyzed (Participants) | 18
events
  AE grade 1 | 18
  AE grade 2 | 7
  AE grade 3 | 1

6. Other Pre Specified Outcome: Number of Participants Able to Perform Self-injections of Peg-interferon
Description: Number of participants able to perform self-injections of peg-interferon.
Time Frame: From initiation of treatment to the first 48 weeks of treatment
Population: 1. subject discontinued treatment after week 1
  2. subjects discontinued treatment after week 12
  1 subject discontinued treatment after week 24
Measure: Count of Participants; unit: Participants
Arm/Group | PegINF-ribavirin
Number analyzed (Participants) | 18
Participants
  Week 0 to Week 12: number analyzed (Participants) | 17
  Week 0 to Week 12: PegINF injected | 17
  Week 0 to Week 12: PegINF not injected | 0
  Week 12 to Week 16: number analyzed (Participants) | 17
  Week 12 to Week 16: PegINF injected | 16
  Week 12 to Week 16: PegINF not injected | 1
  Week 16 to Week 28: number analyzed (Participants) | 15
  Week 16 to Week 28: PegINF injected | 15
  Week 16 to Week 28: PegINF not injected | 0
  Week 28 to Week 32: number analyzed (Participants) | 14
  Week 28 to Week 32: PegINF injected | 13
  Week 28 to Week 32: PegINF not injected | 1
  Week 32 to Week 48: number analyzed (Participants) | 14
  Week 32 to Week 48: PegINF injected | 14
  Week 32 to Week 48: PegINF not injected | 0

7. Other Pre Specified Outcome: Number of Participants With Ribavirin Compliance at ≥ 95%, 80% - 95%, and < 80%
Description: Number of participants with ribavirin compliance at ≥ 95%, 80% - 95%, and < 80%.
Time Frame: From initiation of treatment to the first 48 weeks of treatment
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | PegINF-ribavirin
Number analyzed (Participants) | 18
Participants
  Week 0 to Week 2: number analyzed (Participants) | 17
  Week 0 to Week 2: Compliance < 80% | 0
  Week 0 to Week 2: Compliance 80% - 95% | 2
  Week 0 to Week 2: Compliance ≥ 95% | 15
  Week 2 to Week 4: number analyzed (Participants) | 17
  Week 2 to Week 4: Compliance < 80% | 1
  Week 2 to Week 4: Compliance 80% - 95% | 1
  Week 2 to Week 4: Compliance ≥ 95% | 15
  Week 4 to Week 12: number analyzed (Participants) | 17
  Week 4 to Week 12: Compliance < 80% | 0
  Week 4 to Week 12: Compliance 80% - 95% | 0
  Week 4 to Week 12: Compliance ≥ 95% | 17
  Week 12 to Week 16: number analyzed (Participants) | 17
  Week 12 to Week 16: Compliance < 80% | 0
  Week 12 to Week 16: Compliance 80% - 95% | 1
  Week 12 to Week 16: Compliance ≥ 95% | 16
  Week 16 to Week 20: number analyzed (Participants) | 15
  Week 16 to Week 20: Compliance < 80% | 0
  Week 16 to Week 20: Compliance 80% - 95% | 0
  Week 16 to Week 20: Compliance ≥ 95% | 15
  Week 20 to Week 24: number analyzed (Participants) | 15
  Week 20 to Week 24: Compliance < 80% | 0
  Week 20 to Week 24: Compliance 80% - 95% | 2
  Week 20 to Week 24: Compliance ≥ 95% | 13
  Week 24 to Week 28: number analyzed (Participants) | 15
  Week 24 to Week 28: Compliance < 80% | 1
  Week 24 to Week 28: Compliance 80% - 95% | 0
  Week 24 to Week 28: Compliance ≥ 95% | 14
  Week 28 to Week 32: number analyzed (Participants) | 14
  Week 28 to Week 32: Compliance < 80% | 1
  Week 28 to Week 32: Compliance 80% - 95% | 0
  Week 28 to Week 32: Compliance ≥ 95% | 13
  Week 32 to Week 36: number analyzed (Participants) | 14
  Week 32 to Week 36: Compliance < 80% | 0
  Week 32 to Week 36: Compliance 80% - 95% | 0
  Week 32 to Week 36: Compliance ≥ 95% | 14
  Week 36 to Week 44: number analyzed (Participants) | 14
  Week 36 to Week 44: Compliance < 80% | 0
  Week 36 to Week 44: Compliance 80% - 95% | 1
  Week 36 to Week 44: Compliance ≥ 95% | 13
  Week 44 to Week 48: number analyzed (Participants) | 14
  Week 44 to Week 48: Compliance < 80% | 0
  Week 44 to Week 48: Compliance 80% - 95% | 0
  Week 44 to Week 48: Compliance ≥ 95% | 14

ADVERSE EVENTS:
Time Frame: From enrollment until 6 months after treatment discontinuation
Arm/Group | PegINF-ribavirin
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 2/18
Other Adverse Events (participants affected / at risk) | 13/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PegINF-ribavirin (N=18)
Gastritis (Gastrointestinal disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PegINF-ribavirin (N=18)
Anemia (Blood and lymphatic system disorders) | 8 (9)
Neutropenia (Blood and lymphatic system disorders) | 10 (30)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2014-06-17): https://cdn.clinicaltrials.gov/large-docs/40/NCT02247440/Prot_SAP_ICF_000.pdf